CLINICAL TRIAL: NCT04490252
Title: Effects of Fasting Mimetic Diet on Nephropatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Silvia Lai, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FMD1
Record Dates: First submitted 2020-07-01; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Chronic kidney disease; Fasting mimetic diet; Kidney stem cells
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free diet (No Intervention): Free diet
- FMD (Experimental): Fasting mimetic diet for 5 days, next cycle after 25 days of free diet
  Interventions: Dietary Supplement: Fasting mimetic diet

INTERVENTIONS:
Dietary Supplement: Fasting mimetic diet — Fasting mimetic diet for 5 days, another cycle after 25 days
  Arms: FMD

SUMMARY:
Fasting mimetic diet (FMD) showed positive effects on cardiovascular risks. Purpose of the trial is to evaluate FMD effects on patients affected by chronic kidney disease (CKD), through the stimulation of kidney stem cells and improving cardiovascular and metabolic status.

From April 2018, the investigators enrolled 13 patients (7 male) with an history of primary glomerulonephritis (GMN) and an eGFR between 60 ml/min and 30 ml/min. Exclusion criteria are: age <18 y.o., age> 65 y.o., secondary GMN, severe heart failure (NYHA IV),ongoing infectious diseases, ongoing neoplasia, hepatic diseases, COPD, inflammatory bowel disease, history of stroke, history of acute coronary disease less than 3 months, pregnancy, refuse informed consent.

ELIGIBILITY:
Inclusion Criteria:

* History of primary glomerulonephritis
* eGFR between 60 ml/min and 30 ml/min
* age between 18-65 years old

Exclusion Criteria:

* secondary GMN
* severe heart failure (NYHA IV)
* ongoing infectious diseases
* ongoing neoplasia,
* hepatic diseases
* COPD,
* inflammatory bowel disease
* history of stroke
* history of acute coronary disease less than 3 months
* pregnancy
* refuse informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Blood stem cells level (CD133+, CD24+, CD45-, CD34+, CD309+) (%) | Baseline to 6 months

SECONDARY OUTCOMES:
Creatinine (mg/dl) | Baseline to 6 months
Blood urea (mg/dl) | Baseline to 6 months
Reactive C-protein (mg/L) | Baseline to 6 months
Lipid profile: total cholesterol, LDL, HDL, triglyceride (mg/dl) | Baseline to 6 months
blood glucose (mg/dl) | Baseline to 6 months
iPTH (ng/ml) | Baseline to 6 months
Total protein (g/L) | Baseline to 6 months
Blood insulin (mcUI/ml) | Baseline to 6 months
Blood uric acid (mg/dl) | Baseline to 6 months
Flow-mediated dilation (%) | Baseline to 6 months
Intima-media thickness (mm) | Baseline to 6 months
eGFR using CKD-EPI and MDRD (ml/min/1,73 m2) | Baseline to 6 months
Renal resistive index (dimensionless) | Baseline to 6 months
Epicardial Adipose Tissue (cm) | Baseline to 6 months
Beck depression inventory II (BDI-II) (0 to 63 points) | Baseline to 6 months
BMI (kg/m^2) | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Lai, Prof., Principal Investigator — University of Rome "Sapienza"- Department of Translational and Precision Medicine
Locations (1):
- Hospital "Umberto I", University of Rome "Sapienza", Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No